CLINICAL TRIAL: NCT01804114
Title: Continuous Preperitoneal Infusion of Local Anesthetic Via Pain Pump for Laparoscopic Ventral Hernia Repair
Brief Title: Continuous Local Anesthetic Infusion Following Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Kimberly-Clark Corporation (Industry)
Responsible Party: Principal Investigator, Michael Ujiki MD, Director of Minimally Invasive Surgery, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EH11-297
Record Dates: First submitted 2013-02-25; First posted 2013-03-05 (Estimated); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2020-12

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local anesthetic continuous infusion (Active Comparator): Pain management following hernia repair
  Interventions: Procedure: Pain management following hernia repair
- Placebo continuous infusion (Placebo Comparator): Placebo pain management following hernia repair
  Interventions: Procedure: Placebo for pain management following hernia repair

INTERVENTIONS:
Procedure: Pain management following hernia repair — Continuous infusion of local anesthetic via pain pump following hernia repair
  Other Names: Placement of pain pump to manage post-operative hernia pain
  Arms: Local anesthetic continuous infusion
Procedure: Placebo for pain management following hernia repair — Continuous infusion of placebo via pain pump following hernia repair
  Other Names: Placement of placebo pain pump
  Arms: Placebo continuous infusion

SUMMARY:
The primary endpoint of this study will determine if subjects receiving a continuous infusion of local anesthetic following laparoscopic ventral hernia repair, with the pain pump installed as described to treat post surgical pain will have a lower incidence of pain than those patients treated with a placebo, saline-filled pain pump.The secondary endpoint of this study will determine if subjects receiving a continuous infusion of local anesthetic following laparoscopic ventral hernia repair, with the pain pump installed as described to treat post surgical pain will have a lower utilization of narcotic analgesic medication than those patients treated with the placebo, saline-filled pain pump.

DETAILED DESCRIPTION:
Patients will be screened to determine study eligibility using inclusion/exclusion criteria. Following the consent process, subjects will be randomly assigned to a treatment arm (anesthetic or placebo group). Baseline data will be collected prior surgical implantation of the pain pump delivery system. Both study and control groups will be able to receive supplemental medication for breakthrough pain as determined by the surgeon. Post-operative data will be collected up to three weeks following surgery.

ELIGIBILITY:
Inclusion Criteria:

>18 years

* ASA I,II,III
* Scheduled for Laparoscopic Ventral Hernia Repair

Exclusion Criteria:

* ASA IV or greater
* Needing emergency surgery
* Known history of drug abuse
* GI, liver, kidney or other condition which, per the surgeon's opinion, could interfere with the absorption, distribution, metabolism or excretion of any drug used during the duration of the study
* Patients with a prior allergic reaction or dependency to morphine, demerol, dilaudid, fentanyl, marcaine(bupivicaine), lidocaine, or ropivicaine.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ujiki, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were enrolled and withdrawn prior to assignment of arm/group because their surgeries were converted from laparoscopic to open.
Period: Overall Study
Arm/Group | Local Anesthetic Continuous Infusion | Placebo Continuous Infusion
Started | 17 | 12
Completed | 17 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Anesthetic Continuous Infusion | Placebo Continuous Infusion | Total
Number analyzed (Participants) | 17 | 12 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 8 | 21
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.2) | 60.9 (9.1) | 60.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Post-Operative Pain
Description: Patients will self-report pain assessments on questionnaires each of the first seven days post-operatively using the 4 Point Verbal Rating Scale; ranging from 1=Severe Pain, to 4=No Pain, higher scores indicating less pain, or a better outcome. Values for two daily scores were averaged for each participant, the average across 7 days is reported.
Time Frame: Verbal Rating Scale used twice a day, up to 7 days postoperatively
Population: A verbal rating scale was used to collect self-reported outcomes; higher numbers indicated less pain.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthetic Continuous Infusion | Placebo Continuous Infusion
Number analyzed (Participants) | 17 | 12
score on a scale | 2.91 (.05) | 2.1 (.05)

2. Secondary Outcome: Number of Days With Post-Operative Narcotic Analgesic Use
Description: Patients given a diary to record all narcotics taken post-op for pain control.
Time Frame: Up to 3 weeks post surgery
Population: Subjects recorded days of postoperative narcotics used after discharge (this supplemented pump infusion). Of the total 29 receiving continuous infusion, 13 anesthetic infusion subjects completed the Post Operative Narcotic Analgesic Use Diary, and 8 placebo subjects completed this diary.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Local Anesthetic Continuous Infusion | Placebo Continuous Infusion
Number analyzed (Participants) | 13 | 8
Days | 1 [1 to 4] | 3 [1 to 15]

3. Other Pre Specified Outcome: Satisfaction With PostOperative Pain Management
Description: Subjects report satisfaction with how pain is managed for the first 7 days postoperatively, on a Numerical Rating Scale of 1-10; higher scores indicate less pain and greater satisfaction. Two daily scores were averaged to compute a single value for each day.
Time Frame: Satisfaction scores reported twice daily for up to the 7th day postoperatively
Population: Subjects reported satisfaction of postoperative pain management on a range of 1-10; higher scores indicate less pain and greater satisfaction. The outcome is an average of 7 days of self-reported scores. Of the 17 subjects receiving continuous infusion of local anesthetic, 11 completed this questionnaire, and 6 of the 12 placebo subjects completed this questionnaire.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Local Anesthetic Continuous Infusion | Placebo Continuous Infusion
Number analyzed (Participants) | 11 | 6
units on a scale | 8.3 (.4) | 9 (.5)

ADVERSE EVENTS:
Arm/Group | Local Anesthetic Continuous Infusion | Placebo Continuous Infusion
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/12
Other Adverse Events (participants affected / at risk) | 0/17 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No